CLINICAL TRIAL: NCT01795950
Title: A Phase I Safety and Pharmacodynamic Study of Intravenous Infusion of PLX-PAD Cells in Patients With PAH
Brief Title: Safety Study of PLX-PAD Cells to Treat Pulmonary Arterial Hypertension (PAH)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: United Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PLX-PH-101
Record Dates: First submitted 2013-02-12; First posted 2013-02-21 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: cell therapy; Pulmonary arterial hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 0.5 M PLX-PAD (Experimental): 0.5 million (M) PLX-PAD cells per kg body weight
  Interventions: Drug: PLX-PAD
- 1 M PLX-PAD (Experimental): 1.0 million (M) PLX-PAD cells per kg body weight
  Interventions: Drug: PLX-PAD
- 2 M PLX-PAD (Experimental): 2.0 million (M) PLX-PAD cells per kg body weight
  Interventions: Drug: PLX-PAD

INTERVENTIONS:
Drug: PLX-PAD — intravenous administration of a single dose of PLX-PAD cells
  Other Names: allogeneic Mesenchymal-like Adherent Stromal Cells (ASCs)

SUMMARY:
The purpose of this clinical study is to assess the safety of PLX-PAD to treat pulmonary arterial hypertension (PAH). PLX-PAD is a cell-based product made of allogeneic Mesenchymal-like Adherent Stromal Cells (ASCs), derived from human full-term placentas following an elective caesarean section. This year-long study will evaluate the safety of three different dose levels of PLX-PAD, each given as a single intravenous infusion. This study will also evaluate effects that PLX-PAD may have on PAH, such as changes in the ability to exercise and on other tests used to measure the disease severity.

ELIGIBILITY:
Summary of inclusion and exclusion criteria.

Eligible subjects:

* Are between 18 and 75 years of age
* Have a minimum weight of 45 kg
* Have a diagnosis of idiopathic or heritable PAH, PAH associated with connective tissue disease (CTD), PAH associated with repaired congenital systemic-to-pulmonary cardiac shunt (at least one year since repair), or PAH associated with appetite suppressant/drug or toxin use confirmed by RHC
* Have a current WHO functional class II or III designation
* Have been stabilized, without dose changes for at least 30 days prior to the Screening visit on at least two approved PAH medications (e.g., PDE-5 inhibitor, ERA, prostanoid [as inhalation or infusion]); or IV prostanoid monotherapy. Subjects on an IV prostanoid must have been receiving therapy for at least three months prior to the Screening visit.
* Have a 6MWD equal to or greater than 200 meters (m) at the Screening and Baseline Visits.

Subjects must not:

* Have any evidence of pulmonary thrombus, significant coronary artery disease (CAD), left ventricular dysfunction, or a restrictive or congestive cardiomyopathy
* Have a history of malignancies within the past 5 years,with the exception of individuals with localized, non-metastatic basal cell carcinoma of the skin, in situ carcinoma of the cervix, or prostate cancer who are not currently or expected to undergo radiation therapy, chemotherapy and/or surgical intervention, or to initiate hormonal treatment during the study
* Be listed for transplantation
* Be pregnant or nursing

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-04; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent AEs (frequency and severity at each dose level) | 12 weeks
Incidence of SAEs | 1 year

SECONDARY OUTCOMES:
Change in Six Minute Walk distance | Baseline and 6 weeks
Change in Dyspnea Score | Baseline and 6 weeks
  Change in maximum level of dyspnea experienced during the six minute walk test using a 10 point scale.
Change in WHO Functional Classification | Baseline and 6 weeks
Change in Plasma NT-pro-BNP levels | Baseline and 6 weeks
Change from Baseline in echocardiography parameters | Baseline and 6 weeks
  Change in RV area at end systole and end diastole (for calculation of estimated RV ejection fraction, RV basal and mid diameter at end systole and end diastole, RV free wall thickness, tricuspid annular plane systolic excursion (TAPSE), maximal tricuspid regurgitant jet velocity TRJV) and pulmonary artery end diastolic pressure (PAEDP)
Change in cardiopulmonary hemodynamics | Baseline and 6 weeks
  mean pulmonary arterial pressure (PAPm), heart rate (HR), systolic systemic arterial pressure (SAPs), diastolic systemic arterial pressure (SAPd), mean systemic arterial pressure (SAPm), pulmonary artery systolic pressure (PAPs), pulmonary artery diastolic pressure (PAPd), mean right atrial pressure (RAPm), mean pulmonary capillary wedge pressure (PCWPm), and cardiac output (CO)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Chambers, MRCP FRACP MD, Principal Investigator — The Prince Charles Hospital
Locations (2):
- Australia (2):
  - The Prince Charles Hospital, Brisbane, Queensland
  - The Alfred Hospital, Melbourne